CLINICAL TRIAL: NCT00713089
Title: A 2 Year Prospective Study of Stool Microbiota in Two Diverse Cohorts of Asian (Singaporean and Indonesian) Newborns and Its Influence on Allergy Development
Brief Title: Study of Stool Microbiota in Two Diverse Cohorts of Asian and Its Influence on Allergy Development
Status: Completed | Type: Observational
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Gadjah Mada University (Other)
Responsible Party: Sponsor
Other Study IDs: SQNB01
Record Dates: First submitted 2008-07-07; First posted 2008-07-11 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2014-01

CONDITIONS: Eczema; Asthma; Allergic Rhinitis
Keywords: Eczema; Asthma; Allergic rhinitis; Singapore; Indonesia; Gastrointestinal Flora
MeSH Terms: conditions — Eczema; Asthma; Rhinitis, Allergic

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stools samples will be collected between 72 to 120 hours (or 3 to 5 days) and at 1, 3 and 12 months of age.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: 75 subjects randomised into the placebo arm of an ongoing randomised double-blind placebo controlled clinical trial at National University Hospital, Singapore
- 2: The expecting mothers visiting at the well mother clinics at Gadjah Mada University Hospital were invited to participate in the study

SUMMARY:
This study aims to document prospectively the incidence of allergies of eczema, asthma and allergic rhinitis in 2 diverse cohorts (Singaporean and Indonesian) with contrasting lifestyles and socioeconomic development. The profile of microbial colonization in terms of species variety, as well as their genetic diversity will be studied in Singapore and Indonesia cohorts and to correlate these with clinical allergy.

DETAILED DESCRIPTION:
The main objective of the current study is to establish the relationship of gut microbiota and development of allergy in 2 populations with different socioeconomic status and prevalence of allergy (high in Singapore and low in Indonesia). A cohort of children will be followed prospectively from birth up to 2 years. Stool from different time points, environmental exposure data and clinical manifestations of allergy will be analyzed and recorded. Singapore and Indonesia will provide the South East Asian context in resolving early life influences associated with divergent allergy prevalence. By studying subjects below age two, this will provide valuable knowledge regarding the epidemiology of allergy and atopy in the first years of life, which is poorly documented in this age group. More importantly, the prospective nature and varied parameters included in this study (colony counts, species variety and genetic diversity of microbiota) will add to the global data and scientific evidence for the role of these factors in allergy development.

ELIGIBILITY:
Inclusion Criteria:

* Pre-delivery evaluation

  * Either parent or sibling (ie first degree relative) has a history of atopy. This will be evidenced by a doctor-diagnosis of asthma, allergic rhinitis or eczema AND a positive skin prick test/specific IgE test to any of a panel of common allergens.
  * Parents agree to the child's participation in the study and sign the Informed Consent.
  * The subject and the parents are willing to comply with procedures and both child and parents are able to keep to scheduled clinic visits.
  * Both parents are at contactable range (with valid mobile or land line numbers) for study team to arrange and schedule clinic visits and complete telephone interviews.

Post-delivery evaluation

* The subject is born full term (at least 37 weeks gestation).
* The subject does not have major congenital malformations/major illness as judged by the doctor.
* The subject is in otherwise good, stable health on the basis of medical history, physical examination.
* Family appears to be able to successfully complete this study.

Exclusion Criteria:

* The parent is, in the opinion of the investigator, mentally or legally incapacitated, preventing informed consent from being obtained.
* The parent is unable/ unwilling to comply with procedures.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 75 subjects randomised into the placebo arm of an ongoing randomised double-blind placebo controlled clinical trial at National University Hospital, Singapore.
  For Indonesia Cohort, the expecting mothers visiting at the well mother clinics at Gadjah Mada University Hospital were invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2006-03; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Incidence of allergies of eczema, asthma and allergic rhinitis in 2 diverse cohorts (Singaporean and Indonesian) | 2 years

SECONDARY OUTCOMES:
Gastrointestinal flora in Singapore and Indonesia cohorts | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bee Wah Lee, MD, Principal Investigator — National University Hospital, Singapore
Locations (2):
- Gadjah Mada University Hospital, Yogyakarta, Indonesia
- National University Hospital, Singapore, Singapore